CLINICAL TRIAL: NCT01805362
Title: RAS Blockade at Bedtime Versus on Awakening for the Prevention of Aldosterone Breakthrough
Brief Title: RAS Blockade at Bedtime Versus on Awakening for Aldosterone Breakthrough
Acronym: IRAB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08-API-03
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MORNING (Active Comparator): patients continue to take their treatments (RAS blockers and diuretics) on awaking
  Interventions: Other: Randomization that determine the time of treatment
- EVENING (Experimental): Patients take their treatments(RAS blockers and diurectics)at bedtime
  Interventions: Other: Randomization that determine the time of treatment

INTERVENTIONS:
Other: Randomization that determine the time of treatment
  Other Names: Randomization determine if the treatment will be taken in the morning or in the evening without changing the treatment

SUMMARY:
Objective:

To show that the frequency of aldosterone breakthrough is lower when RAS blockers are given at bedtime compared to on awaking, and to analyze the determinants and consequences of aldosterone breakthrough.

Duration of the study: Inclusion 2 years, follow-up one year, total 3 years Design: prospective, multicenter, randomized, controlled, open label, two parallel groups.

Main selection criteria:

Inclusion criteria

* Chronic kidney disease stage 3 to 4,
* ACEI (captopril, enalapril, or ramipril), and/or ARB (losartan, valsartan, or irbesartan) on awaking for at least three months,
* History of hypertension or proteinuria > 0,5 g/24h or g/g créatininurie.

Exclusion criteria

* Office blood pressure ≥ 160/100 mmHg,
* Anti-aldosterone (spironolactone, eplerenone) or potassium sparing diuretics (modamide, amiloride), or direct renin inhibitor.

Evaluation criteria:

Primary: Serum aldosterone levels at one year.

Secondary:

* Serum aldosterone/renin ratio,
* 24h urine aldosterone,
* Significant aldosterone breakthrough defined by a >10% increase of serum aldosterone levels over baseline values,
* Aldosterone breakthrough defined by an increase of serum aldosterone levels over baseline values,
* HbA1c,
* Urinary albumin/creatinine ratio (UACR) on spot morning urine samples,
* Systolic home blood pressure (SBP),
* Estimated glomerular filtration rate (eGFR) using the MDRD equation.

DETAILED DESCRIPTION:
Rational:

Serum aldosterone levels may increase despite blockade of the renin angiotensin system (RAS) with angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB). This aldosterone breakthrough might be associated with bad outcomes: left ventricular hypertrophy, proteinuria and progression of renal failure. Antihypertensive drugs are given either on awaking or at bedtime. RAS is stimulated during nighttime. RAS blockers and diuretics given on awaking may stimulate aldosterone synthesis, and favor aldosterone breakthrough.

Objective:

To show that the frequency of aldosterone breakthrough is lower when RAS blockers are given at bedtime compared to on awaking, and to analyze the determinants and consequences of aldosterone breakthrough.

Duration of the study: Inclusion 2 years, follow-up one year, total 3 years

Design: prospective, multicenter, randomized, controlled, open label, two parallel groups.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 3 to 4,
* ACEI (captopril, enalapril, or ramipril), and/or ARB (losartan, valsartan, or irbesartan) on awaking for at least three months,
* History of hypertension or proteinuria > 0,5 g/24h or g/g creatininuria,
* Adult with social security insurance,
* Informed consent signed.

Exclusion Criteria:

* Office blood pressure ≥ 160/100 mmHg,
* Pathology with life expectancy < 1 year,
* Anti-aldosterone (spironolactone, eplerenone) or potassium sparing diuretics (modamide, amiloride), or direct renin inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-02-27 (Actual); Primary Completion 2014-04-24 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Serum aldosterone levels at one year | Level change between baseline and one year

SECONDARY OUTCOMES:
Serum aldosterone/renin ratio | level change between baseline and 12 months
Significant aldosterone breakthrough Significant aldosterone breakthrough | changes between baseline and one year
  Significant aldosterone breakthrough defined by a >10% increase of serum aldosterone levels over baseline values,

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ESNAULT, MD, Principal Investigator — Nice University Hospital
Locations (1):
- Department of Nephrology, Nice University Hospital, Nice, France